CLINICAL TRIAL: NCT07248527
Title: PAN-ICIS: Prospective Observational Study Evaluating the Intensive Care Infection Score for Early Detection of Infectious Complications After Pancreatic Resections
Brief Title: PAN-ICIS Study: ICIS for Early Detection of Infectious Complications in Pancreatic Surgery
Acronym: PAN-ICIS
Status: Active, not recruiting | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Štěpán-Ota Schütz, Principal Investigator, Charles University, Czech Republic
Other Study IDs: 108/20-72/2025
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Pancreatectomy; Pancreatic Surgery; Intensive Care (ICU); Inflamatory Markers; Postoperative Care; Postoperative Pancreatic Fistula; Surgical Site Infection After Major Surgery; Postoperative Complications
Keywords: Intensive care infection score; pancreatic surgery; biomarkers; intensive care; sepsis; POPF; Postoperative complications
MeSH Terms: conditions — Postoperative Complications; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients following pancreatic surgery: All patients following pancreatic surgery will be enrolled in this study

SUMMARY:
This study examines a new blood test called ICIS, which may help detect infections earlier after pancreatic surgery. Patients will have routine blood samples taken during their hospital stay, with no extra procedures required. By tracking how ICIS changes over time, investigators aim to improve early infection detection, support safer recovery, and reduce postoperative complications.

DETAILED DESCRIPTION:
Pancreatic resections carry a high burden of postoperative morbidity, particularly due to complications such as pancreatic fistula and bile leakage, which frequently lead to intra-abdominal infection and sepsis. Early diagnosis remains difficult because conventional inflammatory markers (CRP, WBC, PCT, IL-6) lack specificity and are often elevated due to postoperative SIRS. The Intensive Care Infection Score (ICIS) has demonstrated superior performance in distinguishing SIRS from sepsis in surgical patients.

The PAN-ICIS study is a prospective observational study enrolling patients undergoing pancreatic resections. ICIS will be measured postoperatively and compared with conventional inflammatory markers. Perioperative variables, postoperative complications, and infectious outcomes will be collected prospectively. Accurate early differentiation between SIRS and sepsis represents a major need in pancreatic surgery. This study will evaluate the diagnostic accuracy and clinical utility of ICIS for early detection of postoperative infectious complications. If validated, ICIS may support earlier antimicrobial therapy, reduce unnecessary antibiotic exposure, and improve postoperative outcomes in this high-risk population.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18-years-old
* Indication for an elective pancreatic procedure
* Written informed consent

Exclusion Criteria:

* Patients <18 years old.
* Known hematologic malignancy or hematological pathology.
* Refusal to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing pancreatic surgery
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Primary outcome | From day one after surgery to the end of hospitalization
  Diagnostic accuracy of ICIS for detecting postoperative infectious complications, measured by area under the receiver operating characteristic curve (AUROC), sensitivity, specificity, positive and negative predictive values, and likelihood ratios at prespecified cut-offs (e.g., ≥3, ≥4, ≥5).

SECONDARY OUTCOMES:
Secondary outcome | From day one after surgery to the end of the hospitalization
  Comparative diagnostic performance of ICIS vs. CRP, PCT, and IL-6; time-to-diagnosis; and the incremental value of ICIS in multivariable models.

OTHER OUTCOMES:
Exploratory outcomes | From day one after surgery to the end of the 90 day follow-up
  Association of ICIS dynamics with POPF, SSI (superficial/deep/organ-space), bile leak, and anastomotic dehiscence; impact on antibiotic use (duration, de-escalation, escalation) and stewardship metrics; need for radiologic or surgical intervention; length of stay; readmission; and 90-day mortality.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery 2nd Faculty of Medicine, Charles University and Military University Hospital Prague, Prague, Prague 6, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bilimoria KY, Liu Y, Paruch JL, Zhou L, Kmiecik TE, Ko CY, Cohen ME. Development and evaluation of the universal ACS NSQIP surgical risk calculator: a decision aid and informed consent tool for patients and surgeons. J Am Coll Surg. 2013 Nov;217(5):833-42.e1-3. doi: 10.1016/j.jamcollsurg.2013.07.385. Epub 2013 Sep 18. PMID 24055383
- [Background] Cosgrove SE. The relationship between antimicrobial resistance and patient outcomes: mortality, length of hospital stay, and health care costs. Clin Infect Dis. 2006 Jan 15;42 Suppl 2:S82-9. doi: 10.1086/499406. PMID 16355321
- [Background] de Kraker ME, Wolkewitz M, Davey PG, Koller W, Berger J, Nagler J, Icket C, Kalenic S, Horvatic J, Seifert H, Kaasch A, Paniara O, Argyropoulou A, Bompola M, Smyth E, Skally M, Raglio A, Dumpis U, Melbarde Kelmere A, Borg M, Xuereb D, Ghita MC, Noble M, Kolman J, Grabljevec S, Turner D, Lansbury L, Grundmann H. Burden of antimicrobial resistance in European hospitals: excess mortality and length of hospital stay associated with bloodstream infections due to Escherichia coli resistant to third-generation cephalosporins. J Antimicrob Chemother. 2011 Feb;66(2):398-407. doi: 10.1093/jac/dkq412. Epub 2010 Nov 23. PMID 21106563
- [Background] Pierrakos C, Vincent JL. Sepsis biomarkers: a review. Crit Care. 2010;14(1):R15. doi: 10.1186/cc8872. Epub 2010 Feb 9. PMID 20144219
- [Background] Limongelli P, Pai M, Bansi D, Thiallinagram A, Tait P, Jackson J, Habib NA, Williamson RC, Jiao LR. Correlation between preoperative biliary drainage, bile duct contamination, and postoperative outcomes for pancreatic surgery. Surgery. 2007 Sep;142(3):313-8. doi: 10.1016/j.surg.2007.04.022. PMID 17723881
- [Background] Nakamura K, Sho M, Kinoshita S, Akahori T, Nagai M, Nakagawa K, Takagi T, Ikeda N. New insight into the association between bile infection and clinically relevant pancreatic fistula in patients undergoing pancreatoduodenectomy. J Hepatobiliary Pancreat Sci. 2020 Dec;27(12):992-1001. doi: 10.1002/jhbp.781. Epub 2020 Jul 2. PMID 32506812
- [Background] Ohgi K, Sugiura T, Yamamoto Y, Okamura Y, Ito T, Uesaka K. Bacterobilia may trigger the development and severity of pancreatic fistula after pancreatoduodenectomy. Surgery. 2016 Sep;160(3):725-30. doi: 10.1016/j.surg.2016.03.032. Epub 2016 May 24. PMID 27233637
- [Background] Loos M, Strobel O, Legominski M, Dietrich M, Hinz U, Brenner T, Heininger A, Weigand MA, Buchler MW, Hackert T. Postoperative pancreatic fistula: Microbial growth determines outcome. Surgery. 2018 Dec;164(6):1185-1190. doi: 10.1016/j.surg.2018.07.024. Epub 2018 Sep 11. PMID 30217397
- [Background] Droogh DHM, Groen JV, de Boer MGJ, van Prehn J, Putter H, Bonsing BA, van Eijck CHJ, Vahrmeijer AL, van Santvoort HC, Groot Koerkamp B, Mieog JSD. Prolonged antibiotic prophylaxis after pancreatoduodenectomy: systematic review and meta-analysis. Br J Surg. 2023 Oct 10;110(11):1458-1466. doi: 10.1093/bjs/znad213. PMID 37440361
- [Background] Nahm CB, Connor SJ, Samra JS, Mittal A. Postoperative pancreatic fistula: a review of traditional and emerging concepts. Clin Exp Gastroenterol. 2018 Mar 15;11:105-118. doi: 10.2147/CEG.S120217. eCollection 2018. PMID 29588609
- [Background] Saito R, Kawaida H, Amemiya H, Nakata Y, Izumo W, Furuya M, Maruyama S, Takiguchi K, Shoda K, Ashizawa N, Nakayama Y, Shiraishi K, Furuya S, Akaike H, Kawaguchi Y, Ichikawa D. Clinical significance of postoperative complications after pancreatic surgery in time-to-complication and length of postoperative hospital stay: a retrospective study. Langenbecks Arch Surg. 2024 Jun 5;409(1):173. doi: 10.1007/s00423-024-03369-x. PMID 38836878
- [Background] Sankar V, Webster NR. Clinical application of sepsis biomarkers. J Anesth. 2013 Apr;27(2):269-83. doi: 10.1007/s00540-012-1502-7. Epub 2012 Oct 30. PMID 23108494
- [Background] Aloisio E, Dolci A, Panteghini M. Procalcitonin: Between evidence and critical issues. Clin Chim Acta. 2019 Sep;496:7-12. doi: 10.1016/j.cca.2019.06.010. Epub 2019 Jun 10. PMID 31194966
- [Background] Leboueny M, Maloupazoa Siawaya AC, Bouanga LDJ, Mvoundza Ndjindji O, Mveang Nzoghe A, Djoba Siawaya JF. Changes of C-reactive protein and Procalcitonin after four weeks of treatment in patients with pulmonary TB. J Clin Tuberc Other Mycobact Dis. 2023 Jan 18;31:100348. doi: 10.1016/j.jctube.2023.100348. eCollection 2023 May. PMID 36714271
- [Background] Yu CW, Juan LI, Wu MH, Shen CJ, Wu JY, Lee CC. Systematic review and meta-analysis of the diagnostic accuracy of procalcitonin, C-reactive protein and white blood cell count for suspected acute appendicitis. Br J Surg. 2013 Feb;100(3):322-9. doi: 10.1002/bjs.9008. Epub 2012 Nov 30. PMID 23203918
- [Background] Riley LK, Rupert J. Evaluation of Patients with Leukocytosis. Am Fam Physician. 2015 Dec 1;92(11):1004-11. PMID 26760415
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Evans L, Rhodes A, Alhazzani W, Antonelli M, Coopersmith CM, French C, Machado FR, Mcintyre L, Ostermann M, Prescott HC, Schorr C, Simpson S, Wiersinga WJ, Alshamsi F, Angus DC, Arabi Y, Azevedo L, Beale R, Beilman G, Belley-Cote E, Burry L, Cecconi M, Centofanti J, Coz Yataco A, De Waele J, Dellinger RP, Doi K, Du B, Estenssoro E, Ferrer R, Gomersall C, Hodgson C, Moller MH, Iwashyna T, Jacob S, Kleinpell R, Klompas M, Koh Y, Kumar A, Kwizera A, Lobo S, Masur H, McGloughlin S, Mehta S, Mehta Y, Mer M, Nunnally M, Oczkowski S, Osborn T, Papathanassoglou E, Perner A, Puskarich M, Roberts J, Schweickert W, Seckel M, Sevransky J, Sprung CL, Welte T, Zimmerman J, Levy M. Surviving sepsis campaign: international guidelines for management of sepsis and septic shock 2021. Intensive Care Med. 2021 Nov;47(11):1181-1247. doi: 10.1007/s00134-021-06506-y. Epub 2021 Oct 2. No abstract available. PMID 34599691
- [Background] Marchegiani G, Barreto SG, Bannone E, Sarr M, Vollmer CM, Connor S, Falconi M, Besselink MG, Salvia R, Wolfgang CL, Zyromski NJ, Yeo CJ, Adham M, Siriwardena AK, Takaori K, Hilal MA, Loos M, Probst P, Hackert T, Strobel O, Busch ORC, Lillemoe KD, Miao Y, Halloran CM, Werner J, Friess H, Izbicki JR, Bockhorn M, Vashist YK, Conlon K, Passas I, Gianotti L, Del Chiaro M, Schulick RD, Montorsi M, Olah A, Fusai GK, Serrablo A, Zerbi A, Fingerhut A, Andersson R, Padbury R, Dervenis C, Neoptolemos JP, Bassi C, Buchler MW, Shrikhande SV; International Study Group for Pancreatic Surgery. Postpancreatectomy Acute Pancreatitis (PPAP): Definition and Grading From the International Study Group for Pancreatic Surgery (ISGPS). Ann Surg. 2022 Apr 1;275(4):663-672. doi: 10.1097/SLA.0000000000005226. PMID 34596077
- [Background] Quero G, Massimiani G, Lucinato C, Fiorillo C, Menghi R, Laterza V, Schena CA, De Sio D, Rosa F, Papa V, Tortorelli AP, Tondolo V, Alfieri S. Acute pancreatitis after pancreatoduodenectomy: clinical outcomes and predictive factors analysis according to the International Study Group of Pancreatic Surgery definition. HPB (Oxford). 2023 Mar;25(3):363-373. doi: 10.1016/j.hpb.2023.01.002. Epub 2023 Jan 11. PMID 36764909
- [Background] Ho CK, Kleeff J, Friess H, Buchler MW. Complications of pancreatic surgery. HPB (Oxford). 2005;7(2):99-108. doi: 10.1080/13651820510028936. PMID 18333171
- [Background] Aoki S, Miyata H, Konno H, Gotoh M, Motoi F, Kumamaru H, Wakabayashi G, Kakeji Y, Mori M, Seto Y, Unno M. Risk factors of serious postoperative complications after pancreaticoduodenectomy and risk calculators for predicting postoperative complications: a nationwide study of 17,564 patients in Japan. J Hepatobiliary Pancreat Sci. 2017 May;24(5):243-251. doi: 10.1002/jhbp.438. Epub 2017 Apr 5. PMID 28196308
- [Background] Gouma DJ, van Geenen RC, van Gulik TM, de Haan RJ, de Wit LT, Busch OR, Obertop H. Rates of complications and death after pancreaticoduodenectomy: risk factors and the impact of hospital volume. Ann Surg. 2000 Dec;232(6):786-95. doi: 10.1097/00000658-200012000-00007. PMID 11088073
- [Background] Povoski SP, Karpeh MS Jr, Conlon KC, Blumgart LH, Brennan MF. Association of preoperative biliary drainage with postoperative outcome following pancreaticoduodenectomy. Ann Surg. 1999 Aug;230(2):131-42. doi: 10.1097/00000658-199908000-00001. PMID 10450725
- [Background] Kent TS, Sachs TE, Callery MP, Vollmer CM Jr. The burden of infection for elective pancreatic resections. Surgery. 2013 Jan;153(1):86-94. doi: 10.1016/j.surg.2012.03.026. Epub 2012 Jun 13. PMID 22698935
- [Background] Okano K, Hirao T, Unno M, Fujii T, Yoshitomi H, Suzuki S, Satoi S, Takahashi S, Kainuma O, Suzuki Y. Postoperative infectious complications after pancreatic resection. Br J Surg. 2015 Nov;102(12):1551-60. doi: 10.1002/bjs.9919. Epub 2015 Sep 21. PMID 26387569
- [Background] Sourrouille I, Gaujoux S, Lacave G, Bert F, Dokmak S, Belghiti J, Paugam-Burtz C, Sauvanet A. Five days of postoperative antimicrobial therapy decreases infectious complications following pancreaticoduodenectomy in patients at risk for bile contamination. HPB (Oxford). 2013 Jun;15(6):473-80. doi: 10.1111/hpb.12012. Epub 2012 Dec 5. PMID 23458261
- [Background] Smajic J, Tupkovic LR, Husic S, Avdagic SS, Hodzic S, Imamovic S. Systemic Inflammatory Response Syndrome in Surgical Patients. Med Arch. 2018 Apr;72(2):116-119. doi: 10.5455/medarh.2018.72.116-119. PMID 29736100
- [Background] Margraf A, Ludwig N, Zarbock A, Rossaint J. Systemic Inflammatory Response Syndrome After Surgery: Mechanisms and Protection. Anesth Analg. 2020 Dec;131(6):1693-1707. doi: 10.1213/ANE.0000000000005175. PMID 33186158
- [Background] Baddam S, Burns B. Systemic Inflammatory Response Syndrome. 2025 Jun 20. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK547669/ PMID 31613449
- [Background] D'Angelica MI, Ellis RJ, Liu JB, Brajcich BC, Gonen M, Thompson VM, Cohen ME, Seo SK, Zabor EC, Babicky ML, Bentrem DJ, Behrman SW, Bertens KA, Celinski SA, Chan CHF, Dillhoff M, Dixon MEB, Fernandez-Del Castillo C, Gholami S, House MG, Karanicolas PJ, Lavu H, Maithel SK, McAuliffe JC, Ott MJ, Reames BN, Sanford DE, Sarpel U, Scaife CL, Serrano PE, Smith T, Snyder RA, Talamonti MS, Weber SM, Yopp AC, Pitt HA, Ko CY. Piperacillin-Tazobactam Compared With Cefoxitin as Antimicrobial Prophylaxis for Pancreatoduodenectomy: A Randomized Clinical Trial. JAMA. 2023 May 9;329(18):1579-1588. doi: 10.1001/jama.2023.5728. PMID 37078771
- [Background] Vrbacky F, Fatorova I, Blazek M, Smahel P, Zak P. Intensive Care Infection Score (ICIS) is elevated in patients with moderate and severe COVID-19 in the early stages of disease. J Infect Public Health. 2022 May;15(5):533-538. doi: 10.1016/j.jiph.2022.03.018. Epub 2022 Apr 1. PMID 35461075
- [Background] Kaeslin, Martha, Brunner, Saskia, Raths, Janine and Huber, Andreas. "Improvement in detecting bacterial infection in lower respiratory tract infections using the Intensive Care Infection Score (ICIS)" LaboratoriumsMedizin, vol. 40, no. 3, 2016, pp. 175-182.
- [Background] Nierhaus A, Linssen J, Wichmann D, Braune S, Kluge S. Use of a weighted, automated analysis of the differential blood count to differentiate sepsis from non-infectious systemic inflammation: the intensive care infection score (ICIS). Inflamm Allergy Drug Targets. 2012 Apr;11(2):109-15. doi: 10.2174/187152812800392841. PMID 22280231
- [Background] Weimann K, Zimmermann M, Spies CD, Wernecke KD, Vicherek O, Nachtigall I, Tafelski S, Weimann A. Intensive Care Infection Score--A new approach to distinguish between infectious and noninfectious processes in intensive care and medicosurgical patients. J Int Med Res. 2015 Jun;43(3):435-51. doi: 10.1177/0300060514557711. Epub 2015 Apr 7. PMID 25850686
- [Background] van der Geest PJ, Mohseni M, Linssen J, Duran S, de Jonge R, Groeneveld AB. The intensive care infection score - a novel marker for the prediction of infection and its severity. Crit Care. 2016 Jul 7;20(1):180. doi: 10.1186/s13054-016-1366-6. PMID 27384242
- [Background] Deniz E, Klatte S, Tekin-Bubenheim N, Zimmermann M. Intensive care infection score: ICIS discriminates between infected and uninfected critically ill patients in routine intensive care unit practice. Intensive Care Med Exp. 2025 Jun 5;13(1):58. doi: 10.1186/s40635-025-00767-3. PMID 40471473